CLINICAL TRIAL: NCT04177030
Title: Time of Day Effect on Pesticides Metabolism and Toxicity - the CIRCA CHEM Pilot Trial
Brief Title: Time of Day Effect on Pesticides Metabolism and Toxicity
Acronym: CIRCA-CHEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, Konstantinos Makris, Dr. Konstantinos Makris, Associate Professor of Environmental Health, Cyprus University of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CUT3
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diet Habit
Keywords: circadian clock; pesticides; fruits; vegetables; diet; time
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-Morning First (Experimental): Within the first week of the study, Group A will consume fruits and vegetables within time-restriction morning window (9am-12pm). Following washout week, Group A will consume fruits and vegetables within time-restriction night window (7pm-10pm) for one week.
  Interventions: Behavioral: Isopesticide dietary scheme
- Group B-Night First (Experimental): Within the first week of the study, Group B will consume fruits and vegetables within time-restriction night window (7pm-10pm). Following washout week, Group B will consume fruits and vegetables within time-restriction morning window (9am-12pm) for one week.
  Interventions: Behavioral: Isopesticide dietary scheme

INTERVENTIONS:
Behavioral: Isopesticide dietary scheme — All participants should collect first morning urine samples on specific days during the first week and during the third week. Day indicated as "8th", represents the first day of the following week (first day of the wash-out week and first day of the fourth week which is the last day of the study). The participants are asked to consume 4 portions of fruit and 2 portions of vegetables per day during the two trial periods. Overall, dietary daily consumption of foods and fluids will be monitored with the use of a dietary diary throughout the study. Participants will also be asked to take a photograph of the ready to be consumed fruit and vegetable on actual time of consumption and share photos with research team in order to verify at a minimum whether the pre-set time-restriction criteria have been met.
  Other Names: Group A
  Arms: Group A-Morning First
Behavioral: Isopesticide dietary scheme — All participants should collect first morning urine samples on specific days during the first week and during the third week. Day indicated as "8th", represents the first day of the following week (first day of the wash-out week and first day of the fourth week which is the last day of the study). The participants are asked to consume 4 portions of fruit and 2 portions of vegetables per day during the two trial periods. Overall, dietary daily consumption of foods and fluids will be monitored with the use of a dietary diary throughout the study. Participants will also be asked to take a photograph of the ready to be consumed fruit and vegetable on actual time of consumption and share photos with research team in order to verify at a minimum whether the pre-set time-restriction criteria have been met.
  Other Names: Group B
  Arms: Group B-Night First

SUMMARY:
The CIRCA-CHEM study is a non-pharmacological, randomized cross-over health intervention trial studying the effect of the time of day on the metabolism and concomitant toxicity of exposures to pesticides found in a balanced fruits and vegetables diet, providing the same weekly portions of fruit and vegetables (isopesticide dietary scheme) but consumed in two different time windows (morning vs. night).

DETAILED DESCRIPTION:
The investigator's study is a 2x2 randomized cross over trial. All participants will be randomly allocated to one of the two groups (morning vs night or night first and then morning; Groups A and B, respectively) having to daily consume an isopesticide dietary pattern (4:2 portions of fruits:vegetables) within a specific, time-restricted window for a week and repeat the same procedure within a different time-restricted window for another week after an in between wash-out period of one week. Morning time-restriction window is set to be between 9am until 12pm and nighttime-restriction window is set between 7pm until 10pm, respectively. Participants will be called to start time-restriction based on group allocation.

In order for all participants to enter the study at a baseline level of pesticide load they will be asked to undergo a run-in day where no fruit and vegetable consumption is allowed prior the onset of the study. Within the first week of the study, Group A (n=25) will consume fruits and vegetables within time-restriction morning window (9am-12pm) and Group B (n=25) will consume fruits and vegetables within time-restriction night window (7pm-10pm). After washout week period where participants will be called to return to their usual dietary habits, two groups will swap to the opposite time-restriction window.

All participants should collect first morning urine samples on specific days during the first week (1st, 3rd, 5th, 8th day) and during the third week (1st, 3rd, 5th, 8th day). Day indicated as "8th", represents the first day of the following week (first day of the wash-out week and first day of the fourth week which is the last day of the study). The participants are asked to consume 4 portions of fruit and 2 portions of vegetables per day during the two trial periods. The fruits selected for the study that will take place during winter season of 2020 are: a pear (~180g), a red apple (~170g), a banana (~110g) and an orange (~400g). The vegetables selected include a tomato (~200g), two cucumbers (~240g) and lettuce (1 cup,4 chopped). All fruits and vegetables will be freshly and seasonally produced in Cyprus. Overall, dietary daily consumption of foods and fluids will be monitored with the use of a dietary diary throughout the study. Participants will also be asked to take a photograph of the ready to be consumed fruit and vegetable on actual time of consumption and share photos with research team in order to verify at a minimum whether the pre-set time-restriction criteria have been met.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults (absence of any self-reported chronic or other known disease)
2. Age:18-60
3. Normal to overweight individuals (18.5 ≤ BMI <30)
4. Permanent residents of Cyprus for the past 5 years

Exclusion Criteria:

1. Chronically ill individuals (subjects with no self-reported chronic diseases)
2. Age <18 years
3. Obese individuals (BMI ≥30)
4. Pregnant or lactating women
5. Individuals with food allergies
6. Systematic organic consuming individuals (more than 80% of their weekly meals)
7. Individuals working shift schedule or having chronic sleep symptoms

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in concentrations of biomarkers of exposure to pesticides (ng/g) from baseline | up to day 8 in both periods since baseline
  pyrethroids and neonicotinoids urinary levels in each period
Change in peak area counts of the metabolomic profile from baseline | up to day 8 in both periods since baseline
  the metabolomic profile in each period using a metabolomics platform

SECONDARY OUTCOMES:
Change in levels of weight in kilograms | up to day 8 in both periods since baseline
  weight measurements
Change in levels of waist circumference in centimeters | up to day 8 in both periods since baseline
  waist circumference measurements

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos C Makris, Principal Investigator — Cyprus University of Technology
Locations (1):
- Cyprus University of Technology, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Upon publication the individual participant data (in anonymized form) will be available through the journal's website.
Time Frame: upon publication, the data will become available.
Access Criteria: the data will be publicly available